CLINICAL TRIAL: NCT05095831
Title: Endoscopic Ultrasound Shear Wave for Neoplasia and Inflammation Assessment Among Solid Pancreas Lesions: a Case-control Observational Trial.
Brief Title: EUS Shear Wave for Solid Pancreatic Lesions.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: IECED-10152021
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Pancreas Neoplasm; Pancreatitis; Pancreatitis, Acute; Pancreatitis, Chronic; Pancreatitis, Autoimmune
Keywords: Pancreatic Neoplasms; Carcinoma, Pancreatic Ductal; Pancreatic Intraductal Neoplasms; Pancreatitis; Pancreatitis, Chronic; Pancreatitis, Alcoholic; Pancreatitis, Acute Necrotizing; Pancreatitis, Acute Hemorrhagic; Autoimmune Pancreatitis
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis; Pancreatitis, Chronic; Autoimmune Pancreatitis; Carcinoma, Pancreatic Ductal; Pancreatic Intraductal Neoplasms; Pancreatitis, Alcoholic; Pancreatitis, Acute Necrotizing; Pancreatitis, Acute Hemorrhagic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Suspicion of solid neoplastic lesion: Patients with high suspicion of solid pancreas neoplasia: carcinoma, intrapapillary mucinous neoplasia (IPMN), neuroendocrine tumor, lymphoma, or intrapancreatic metastasis; based on CT/MR.
  Interventions: Diagnostic Test: Pancreas EUS shear wave; Diagnostic Test: Pancreas EUS-elastography and EUS-guided biopsy
- Suspicion of a solid inflammatory lesion: Patients with high suspicion of solid inflammatory lesions: acute, chronic, or autoimmune pancreatitis; based on CT/MR.
  Interventions: Diagnostic Test: Pancreas EUS shear wave; Diagnostic Test: Pancreas EUS-elastography and EUS-guided biopsy
- Control group: Patients without a history of any type of solid or hematologic malignancy, hepato-pancreato-biliary disease (including fatty liver and pancreas disease), tobacco/alcohol habits, or morbid obesity with bariatric surgery criteria; who require EUS evaluation (e.g., suspicious of a subepithelial lesion in the context of chronic dyspepsia).
  Interventions: Diagnostic Test: Pancreas EUS shear wave; Diagnostic Test: Pancreas EUS-elastography and EUS-guided biopsy

INTERVENTIONS:
Diagnostic Test: Pancreas EUS shear wave — EUS Shear wave elastography (SWE) is a form of ultrasound elastography used in transabdominal ultrasonography. It measures tissue elasticity by generating shear waves inside the organ using the acoustic radiation force impulse (ARFI). The ultrasound machine monitors shear wave propagation and measures the velocity. The shear wave velocity, displayed in kilopascals [kPa] or meters per second. Also, the dispersion slope or ultrasound shear wave dispersion (SWD) will be recorded. It is the measure of viscosity [(m/sec)/kHz] using SWE.
  A first endoscopist will perform EUS over pancreas tissue. Without any elastography assessment (strain ratio/histogram) , the endoscopist will take ten shear wave measurements of pancreas tissue elasticity by generating shear waves inside the pancreas using the ARFI.
Diagnostic Test: Pancreas EUS-elastography and EUS-guided biopsy — Pancreas EUS-elastography measures the pancreatic tissue stiffness through strain ratio (SR) and strain histogram (SH).
  A second endoscopist blind to pancreas tissue shear wave findings will perform EUS-elastography with corresponding SR and SH measurements. The SR/SH will be measured and documented. Finally, a pancreas tissue biopsy will be performed. The impossibility of biopsy is an exclusion criterion (except in control patients). Due to ethical purposes, a biopsy will not be performed on patients from the control group.

SUMMARY:
The diagnosis of pancreas diseases is based on a combination of clinical signs, symptoms, and laboratory tests, but mainly on imaging techniques such as computed tomography (CT) and magnetic resonance (MR). However, CT/MR have variable sensitivity and specificity, with certain disadvantages. Endoscopic ultrasound with elastography is an important resource with higher diagnostic accuracy in assessing solid pancreas lesions. Shear wave velocities of healthy parenchyma, acute, chronic and autoimmune pancreatitis, neoplastic lesions of the pancreas must be evaluated and compared.

DETAILED DESCRIPTION:
The pancreas is a retroperitoneal organ that can cause inflammatory and neoplastic diseases, significantly impacting the quality of life to survival. Acute pancreatitis is one of the most frequent gastrointestinal causes for hospital admission in industrialized countries. Chronic pancreatitis, although lower in incidence, significantly reduces patients' quality of life. Pancreas cancer is one of the neoplastic diseases with high mortality worldwide. Those diseases have been associated with significant morbidity, mortality, and hospitalization costs

The diagnosis of pancreas diseases is based on a combination of clinical signs, symptoms, and laboratory tests, but mainly on imaging techniques such as computed tomography (CT) and magnetic resonance (MR). Imaging provides a significant contribution to the diagnosis of pancreatic diseases and severity estimation or staging for inflammatory and neoplastic lesions, respectively. However, CT/MR have variable sensitivity and specificity, with certain disadvantages.

Endoscopic ultrasound with elastography is an important resource with higher diagnostic accuracy in assessing solid pancreas lesions. Shear wave elastography is a novel technique that can measure tissue elasticity by generating shear waves inside the organ using the acoustic radiation force impulse.

EUS Shear wave velocities of healthy parenchyma and solid pancreas lesions as acute, chronic, autoimmune pancreatitis and neoplasia are under described and must be evaluated and contrasted. Therefore, the present study pursues to estimate the diagnostic accuracy of EUS Shear wave for neoplasia assessment among solid pancreas lesions.

ELIGIBILITY:
Inclusion Criteria:

* Neoplasia group: high suspicion of pancreas neoplasia based on computed tomography and/or nuclear magnetic resonance.
* Inflammatory group: high suspicion of acute or chronic pancreatitis based on computed tomography and/or nuclear magnetic resonance.
* Control group: patients without a history of any type of solid or hematologic malignancy, hepato-pancreato-biliary disease (including fatty liver and pancreas disease), tobacco/alcohol habits, or morbid obesity with bariatric surgery criteria; who require EUS evaluation (e.g., suspicious of a subepithelial lesion in the context of chronic dyspepsia).

Exclusion Criteria:

* Uncontrolled coagulopathy, kidney/liver failure, or any comorbidity with important impact on cardiac risk assessment (NHYA III/IV);
* Impossibility of EUS-guided biopsy (only for neoplasia or inflammatory group);
* Pregnancy or nursing;
* Refuse to participate in the study and/or to sign corresponding informed consent.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with solid pancreas lesions with an indication of EUS assessment.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
SWE/SWD pancreas EUS shear wave | Two months
  The median of ten SWE/SWD measures will be calculated to represent the final pancreas tissue shear wave measure per case. The higher the median, the more suspicious for neoplasia.
SR/SH pancreas EUS-elastography | Two months
  The SR/SH measures will be recorded per case. A SR>15 kPa and a SH≤45 will be considered as highly suspicious for neoplasia.
EUS-biopsied histopathology findings | One month
  The pathologist will have access to all the clinical data of each patient, including EUS-elastography findings, except shear wave measurements, to determine if the assessed pancreas lesion was neoplasia or inflammatory. In addition, a preliminary diagnostic accuracy (sensitivity, specificity, positive and negative predictive value) of pancreas EUS shear wave measurements and pancreas EUS-elastography will be calculated using histopathology results as gold standard.
Clinical condition at one-year follow-up | One year
  A gastroenterologist will follow patients for one year after the procedure. During this follow-up, there will record cases who undergo exploratory or onco-specific surgery (histopathology) and the number of patients who undergo onco-specific treatment (radiotherapy, radiosurgery, chemotherapy, and biological therapy) or clinical management/surveillance. Survival and cause of death will also be recorded when corresponding. This follow-up purposes of determining definitively if the assessed pancreas lesion was neoplasia or inflammatory. A definitive diagnostic accuracy (sensitivity, specificity, positive and negative predictive value) of pancreas EUS shear wave measurements and pancreas EUS-elastography will be calculated using a one-year follow-up as the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MD FASGE, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Okasha H, Elkholy S, El-Sayed R, Wifi MN, El-Nady M, El-Nabawi W, El-Dayem WA, Radwan MI, Farag A, El-Sherif Y, Al-Gemeie E, Salman A, El-Sherbiny M, El-Mazny A, Mahdy RE. Real time endoscopic ultrasound elastography and strain ratio in the diagnosis of solid pancreatic lesions. World J Gastroenterol. 2017 Aug 28;23(32):5962-5968. doi: 10.3748/wjg.v23.i32.5962. PMID 28932088
- [Result] Bayramoglu Z, Akyol Sari ZN, Koker O, Adaletli I, Eker Omeroglu R. Shear wave elastography evaluation of liver, pancreas, spleen and kidneys in patients with familial mediterranean fever and amyloidosis. Br J Radiol. 2021 Dec;94(1128):20210237. doi: 10.1259/bjr.20210237. Epub 2021 Sep 14. PMID 34520686
- [Result] Platz Batista da Silva N, Engesser M, Hackl C, Brunner S, Hornung M, Schlitt HJ, Evert K, Stroszczynski C, Jung EM. Intraoperative Characterization of Pancreatic Tumors Using Contrast-Enhanced Ultrasound and Shear Wave Elastography for Optimization of Surgical Strategies. J Ultrasound Med. 2021 Aug;40(8):1613-1625. doi: 10.1002/jum.15545. Epub 2020 Oct 30. PMID 33124700
- [Result] Suzuki H, Ishikawa T, Ohno E, Iida T, Uetsuki K, Yashika J, Yamada K, Yoshikawa M, Furukawa K, Nakamura M, Honda T, Ishigami M, Kawashima H, Fujishiro M. An initial trial of quantitative evaluation of autoimmune pancreatitis using shear wave elastography and shear wave dispersion in transabdominal ultrasound. Pancreatology. 2021 Jun;21(4):682-687. doi: 10.1016/j.pan.2021.02.014. Epub 2021 Feb 20. PMID 33648879